CLINICAL TRIAL: NCT06239766
Title: Assessing Breast Cancer Risk Prior to Gender-Affirming Chest Masculinization Surgery in Transgender and Gender-Diverse Persons
Brief Title: BC Risk Assessment Before Top Surgery
Status: Completed | Type: Observational
Sponsor: Medical College of Wisconsin (Other)
Responsible Party: Principal Investigator, Chandler S Cortina, Assistant Professor of Surgery, Medical College of Wisconsin
Other Study IDs: PRO00045830
Record Dates: First submitted 2024-01-16; First posted 2024-02-02 (Actual); Last update posted 2024-03-13 (Actual); Status verified 2024-03

CONDITIONS: Breast Cancer; Risk Reduction
Keywords: Transgender; Gender Diverse; Nonbinary; Risk Assessment; Mastectomy; Top Surgery
MeSH Terms: conditions — Breast Neoplasms; Risk Reduction Behavior

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Non-Cisgender Adults Considering Chest Masculinization Surgery: Persons assigned female or intersex at birth who identify as TGD and are considering gender-affirming chest masculinization surgery.
  Interventions: Diagnostic Test: Breast Cancer Risk Assessment

INTERVENTIONS:
Diagnostic Test: Breast Cancer Risk Assessment — Gail and IBIS Tools will be utilized to calculate mean lifetime breast cancer risk

SUMMARY:
The population of transgender and gender-diverse (TGD) persons in Wisconsin and the U.S. is steadily increasing. As this population grows, the number of individuals seeking gender-affirming therapies, including gender-affirming operations and gender-affirming hormone therapy, is also growing. An example of gender-affirming surgery is chest masculinization surgery, in which most breast tissue is removed in a person assigned female or intersex at birth to allow the chest to appear masculine. Gender-affirming chest masculinization surgery is not generally considered equivalent to an oncologic mastectomy, which aims to removal all breast tissue for future breast cancer reduction or current breast cancer treatment.

The goals of this investigation are to 1) determine the percent of TGD persons considering chest masculinization surgery who have an elevated lifetime risk of breast cancer development and/or a pathogenic genetic mutation; 2) measure the percent who are at risk and choose to undergo risk-reducing mastectomies as part of chest masculinization surgery; and 3) assess and compare self-perceived breast cancer risk with calculated risk.

The results of this study will substantially inform TGD patients and surgeons on the utility of personalized breast cancer risk assessment prior to chest masculinization surgery and the accuracy of self-perceived breast cancer risk in TGD persons.

ELIGIBILITY:
Inclusion Criteria:

1. ≥18 years old.
2. Assigned female or intersex at birth and identify as non-cisgender.
3. Any individual considering undergoing gender-affirming chest masculinization surgery
4. Ability to communicate in English.
5. Ability to understand a written informed consent document, and the willingness to sign it.

Exclusion Criteria:

1. <18 years old.
2. Assigned male sex at birth.
3. Previously underwent chest masculinization surgery or any form of oncological mastectomy for the purposes of risk-reduction or cancer treatment.
4. Any previous or current history of breast cancer, including ductal carcina in situ (DCIS).
5. Inability to communicate in English.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Persons who identify as transgender, nonbinary, and/or gender-diverse (TGD) who were assigned female and/or intersex at birth.
Study Population: TGD persons considering chest masculinization surgery.
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2023-03-15 (Actual); Primary Completion 2023-12-29 (Actual); Study Completion 2024-02-01 (Actual)

PRIMARY OUTCOMES:
Estimated prevalence of TGD persons seeking chest masculinization surgery who at an elevated breast cancer risk. | 1 year
  Validated breast cancer risk calculators (IBIS and Gail) will be used to determine lifetime breast cancer risk of participants enrolled into the study. Ranges and 95% CI will be made to estimate the percent of TGD persons at risk.
Rate of uptake of oncologic risk reducing mastectomies as part of chest masculinization surgery in TGD persons at risk of breast cancer based on validated models. | 1 year
  To determine whether those TGD persons at elevated risk of breast cancer development choose to undergo risk-reducing mastectomies as part of their chest masculinization surgery.
Self-perceived breast cancer risk vs calculated breast cancer risk | 1 year
  A visual analog scale from 0-100% will be used to compare and assess the self-perceived estimated breast cancer risk with calculated breast cancer risk. 13% is marked as the average cisgender women's risk of breast cancer and participants report their self-perceived risk as single whole integer (ex. 8%, 15%, 25%, etc.) on the scale from 0-100% where 0-12% represents below average risk person and 13-100% represent above average risk.

CONTACTS AND LOCATIONS:
Overall Officials: Chandler S Cortina, Principal Investigator — The Medical College of Wisconsin
Locations (1):
- Medical College of Wisconsin, Milwaukee, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cortina CS. ASO Author Reflections: A Breast Cancer Risk Assessment and the Decision for Gender-Affirming Chest Masculinization Surgery or Oncologic Risk-Reducing Mastectomies in Transgender and Gender-Diverse Individuals. Ann Surg Oncol. 2024 Oct;31(11):7483-7484. doi: 10.1245/s10434-024-15801-z. Epub 2024 Jul 26. No abstract available. PMID 39060689
- [Derived] Cortina CS, Purdy A, Brazauskas R, Stachowiak SM, Fodrocy J, Klement KA, Sasor SE, Krucoff KB, Robertson K, Buth J, Lakatos AEB, Petroll AE, Doren EL. The Impact of a Breast Cancer Risk Assessment on the Decision for Gender-Affirming Chest Masculinization Surgery in Transgender and Gender-Diverse Individuals: A Pilot Single-Arm Educational Intervention Trial. Ann Surg Oncol. 2024 Oct;31(11):7474-7482. doi: 10.1245/s10434-024-15701-2. Epub 2024 Jun 28. PMID 38940898

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-01-30): https://cdn.clinicaltrials.gov/large-docs/66/NCT06239766/Prot_SAP_000.pdf
  • Informed Consent Form (2023-02-20): https://cdn.clinicaltrials.gov/large-docs/66/NCT06239766/ICF_001.pdf